CLINICAL TRIAL: NCT07013175
Title: WIse CHoices in the Intensive Care Unit, a Cluster Randomized Registry Based Clinical Trial
Brief Title: Wise Choices in the Intensive Care Unit
Acronym: WICH-ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Uppsala-Örebro Regional Research Council (Other); Vastra Gotaland Region (Other Government); Region Jönköping County (Other Government); Region Skane (Other); Region Stockholm (Other Government); Sormland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Max Bell, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WICH-ICU
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Critical Illness; Ventilation; Outcome; Dialysis; Acute Kidney Injury
Keywords: critical illness; choosing wisely
MeSH Terms: conditions — Critical Illness; Respiratory Aspiration; Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: There are two phases in this block randomized stepped-wedge ICU study, the control phase and the intervention phase. All participating ICU's start with a control period. During this phase, clinical monitors assess the number of arterial blood gases, -venous tests and number of chest x-rays performed at the ICU. This monitoring will assess all patients treated during a week and report tests per patient per day. As ICU's are randomized to the intervention phase the same clinical monitoring will be performed. Importantly, after six- and 12 months (irrespective of randomization allocation, if the ICU is still in the control- or intervention phase), the clinical monitor will re-assess the testing/diagnostic metrics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Choosing wisely intervention (Active Comparator): The Choosing Wisely (CW) protocol in the critical care setting; specifically minimizing the number of arterial blood gases, number of venous tests and number of chest x-rays
  Interventions: Procedure: Choosing wisely protocol
- Choosing wisely control (No Intervention): Regular critical care

INTERVENTIONS:
Procedure: Choosing wisely protocol — Se arm description
  Arms: Choosing wisely intervention

SUMMARY:
Aim: to evaluate if the Choosing Wisely campaign can be introduced without harming critically ill patients.

Background: Each year, around 45,000 patients are admitted to Sweden's 81 ICUs (intensive care units), costing 6-7 billion SEK (6% of total healthcare expenditure). The high costs of health care are partly attributable to overuse of diagnostic tests. Up to 30% of these tests lead to treatments that provide no benefit for patients, some of them may even be harmful(1-3). To improve quality of care while combating this problem of cost, the American Board of Internal Medicine Foundation developed the Choosing Wisely Campaign, tasking professional societies to develop lists of top five medical services patients and physicians should question. Patients in the ICU, can especially benefit from this paradigm shift. They are subjected to multiple testing on a daily - sometimes hourly - basis, therefore this field of medicine responded to the campaign quickly. Two sets of top-five-lists of tests and interventions that can be questioned have been published(4 5).

In multiple countries, including Sweden, the Choosing Wisely campaign is gathering traction among critical care physicians and is on the verge of being introduced. It is both common-sensical and will save money, so health care leaders are positive. However, the investigators have an opportunity, and a duty, to assess the evidence; can the Choosing Wisely campaign be introduced without harming ICU patients?

The present study thus aims to evaluate the introduction of the Choosing Wisely campaign in the context of the ICU. Is this change of care strategy associated with changes in 30-day-mortality? Secondary outcomes include ICU length of stay, use of non-invasive- or invasive mechanical ventilation and continuous renal replacement therapy. This is a registry-based cluster randomized controlled study (R-RCT), targeting Swedish ICU's across multiple regions. Primary and secondary outcomes will be retrieved from the Swedish Intensive care Register (SIR), making ICU participation easier and less costly.

DETAILED DESCRIPTION:
Purpose and aims Aim: to evaluate if the Choosing Wisely campaign can be introduced without harming critically ill patients.

Background: Each year, around 45,000 patients are admitted to Sweden's 81 ICUs (intensive care units), costing 6-7 billion SEK (6% of total healthcare expenditure). The high costs of health care are partly attributable to overuse of diagnostic tests. Up to 30% of these tests lead to treatments that provide no benefit for patients, some of them may even be harmful. To improve quality of care while combating this problem of cost, the American Board of Internal Medicine Foundation developed the Choosing Wisely Campaign, tasking professional societies to develop lists of top five medical services patients and physicians should question. Patients in the ICU, can especially benefit from this paradigm shift. They are subjected to multiple testing on a daily - sometimes hourly - basis, therefore this field of medicine responded to the campaign quickly. Two sets of top-five-lists of tests and interventions that can be questioned have been published.

In multiple countries, including Sweden, the Choosing Wisely campaign is gathering traction among critical care physicians and is on the verge of being introduced. It is both common-sensical and will save money, so health care leaders are positive. However, the investigators have an opportunity, and a duty, to assess the evidence; can the Choosing Wisely campaign be introduced without harming ICU patients?

The present study thus aims to evaluate the introduction of the Choosing Wisely campaign in the context of the ICU. Is this change of care strategy associated with changes in 30-day-mortality? Secondary outcomes include ICU length of stay, use of non-invasive- or invasive mechanical ventilation and continuous renal replacement therapy as well as unplanned readmissions. This is a registry-based cluster randomized controlled study (R-RCT), targeting Swedish ICU's across multiple regions. Primary and secondary outcomes will be retrieved from the Swedish Intensive care Register (SIR), making ICU participation easier and less costly.

Survey of the field Investigations on mortality, ICU length of stay (LOS) or effect on organ support among critically ill patients after the introduction of the Choosing Wisely protocol are lacking. Evidence suggests that routine laboratory testing is associated with preventable harms, such as hospital-acquired anemia and further unnecessary testing.

Can ICUs reduce unnecessary diagnostics? A Canadian single center before- and after study aimed at reducing (unnecessary diagnostic) phlebotomy in the ICU. They showed a decrease of 6.6mL/patient-day, blood tube consumption decreased, amounting to 13276 tubes saved over 11 months. Red blood cell transfusions decreased significantly.

Study design Research questions Can the Choosing Wisely protocol, specifically minimizing the number of arterial blood gases, -venous tests and -chest x-rays, be introduced safely in Swedish ICU's?

P: Adult patients treated in Swedish intensive care units.

I: The Choosing Wisely (CW) protocol, specifically minimizing the number of arterial blood gases, number of venous tests and number of chest x-rays

C: ICU care as of today, without the introduction of the CW protocol. Each ICU is its own and others' control.

O: Primary outcome: 30-day-mortality. Secondary outcomes: ICU length of stay, time in invasive/ non-invasive mechanical ventilation, time on continuous renal replacement therapy and unplanned readmissions within 72 hours of ICU discharge.

Variables and measures There are two phases in this block randomized stepped-wedge ICU study, the control phase and the intervention phase. All participating ICU's start with a control period. During this phase, clinical monitors assess the number of arterial blood gases, -venous tests and number of chest x-rays performed at the ICU. This monitoring will assess all patients treated during a week and report tests per patient per day. As ICU's are randomized to the intervention phase the same clinical monitoring will be performed. Importantly, after six- and 12 months (irrespective of randomization allocation, if the ICU is still in the control- or intervention phase), the clinical monitor will re-assess the testing/diagnostic metrics.

Outcomes from this R-RCT will be extracted using the Swedish Intensive care Register (SIR). These include the primary outcome, 30-day-mortality and secondary outcomes: ICU length of stay, time in invasive/non-invasive mechanical ventilation, time on continuous renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older, treated in Swedish ICU's

Exclusion Criteria:

* Patients under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days after index ICU admission
  Death within 30 days of ICU admission

SECONDARY OUTCOMES:
ICU length of stay | Up to one year after index ICU admission
  Days in the ICU after index ICU admission
Time in invasive/ non-invasive mechanical ventilation | Up to one year after index ICU admission
  Days in the ICU in invasive or non-invasive mechanical ventilation
Time on continuous renal replacement therapy | Up to one year after index ICU admission
  Days in the ICU on continuous renal replacement therapy
ICU readmission | 72 hours post ICU discharge
  Unplanned ICU readmission within 72h of ICU discharge

OTHER OUTCOMES:
ICU readmission | Within 72 hours of ICU discharge
  Readmissions after ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Max B Bell, MD, PhD, Principal Investigator — N32276 PMI/Karolinska
Locations (2):
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Karolinska Institutet, Stockholm

IPD SHARING:
Plan to Share IPD: No
This study uses data on a block level from participating ICUs; therefore it is not feasible to share IPD, but we may opt to share other information

REFERENCES:
- [Background] Costante A, Chen XK, Dudevich A, Dennis Christy A, Francis L, Chui C. Overuse of Tests and Treatments: Has Canada Made Progress? Healthc Q. 2023 Jan;25(4):10-12. doi: 10.12927/hcq.2023.27024. PMID 36826234
- [Background] Mafi JN, Reid RO, Baseman LH, Hickey S, Totten M, Agniel D, Fendrick AM, Sarkisian C, Damberg CL. Trends in Low-Value Health Service Use and Spending in the US Medicare Fee-for-Service Program, 2014-2018. JAMA Netw Open. 2021 Feb 1;4(2):e2037328. doi: 10.1001/jamanetworkopen.2020.37328. PMID 33591365
- [Background] Shrank WH, Rogstad TL, Parekh N. Waste in the US Health Care System: Estimated Costs and Potential for Savings. JAMA. 2019 Oct 15;322(15):1501-1509. doi: 10.1001/jama.2019.13978. PMID 31589283
- [Background] Halpern SD, Becker D, Curtis JR, Fowler R, Hyzy R, Kaplan LJ, Rawat N, Sessler CN, Wunsch H, Kahn JM; Choosing Wisely Taskforce; American Thoracic Society; American Association of Critical-Care Nurses; Society of Critical Care Medicine. An official American Thoracic Society/American Association of Critical-Care Nurses/American College of Chest Physicians/Society of Critical Care Medicine policy statement: the Choosing Wisely(R) Top 5 list in Critical Care Medicine. Am J Respir Crit Care Med. 2014 Oct 1;190(7):818-26. doi: 10.1164/rccm.201407-1317ST. PMID 25271745
- [Background] Zimmerman JJ, Harmon LA, Smithburger PL, Chaykosky D, Heffner AC, Hravnak M, Kane JM, Kayser JB, Lane-Fall MB, Matos RI, Mauricio RV, Murphy DJ, Nurok M, Reddy AJ, Ringle E, Seferian EG, Smalls-Mantey NM, To KB, Kaplan LJ. Choosing Wisely For Critical Care: The Next Five. Crit Care Med. 2021 Mar 1;49(3):472-481. doi: 10.1097/CCM.0000000000004876. PMID 33555779
- [Background] Salisbury AC, Reid KJ, Alexander KP, Masoudi FA, Lai SM, Chan PS, Bach RG, Wang TY, Spertus JA, Kosiborod M. Diagnostic blood loss from phlebotomy and hospital-acquired anemia during acute myocardial infarction. Arch Intern Med. 2011 Oct 10;171(18):1646-53. doi: 10.1001/archinternmed.2011.361. Epub 2011 Aug 8. PMID 21824940
- [Background] Bodley T, Levi O, Chan M, Friedrich JO, Hicks LK. Reducing unnecessary diagnostic phlebotomy in intensive care: a prospective quality improvement intervention. BMJ Qual Saf. 2023 Aug;32(8):485-494. doi: 10.1136/bmjqs-2022-015358. Epub 2023 Jan 19. PMID 36657786